CLINICAL TRIAL: NCT03167320
Title: Low Von Willebrand in Ireland Cohort Study
Acronym: LOVIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, James O'Donnell, George Gabriel Stokes Professor of Haematology, Director Haemostasis Research Group, St. James's Hospital, Ireland
Other Study IDs: LOVIC01
Record Dates: First submitted 2016-04-06; First posted 2017-05-25 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Von Willebrand Factor, Deficiency
MeSH Terms: conditions — Von willebrand factor, deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood samples will be taken at study enrolment and stored for further analysis, including samples for DNA analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LOVIC: Irish patients with low Von Willebrand levels will be have both venous blood sampling and a bleeding score administered at study entry. A DDAVP (1-desamino-8-D-arginine vasopressin) fall off study was organised for those patients in the cohort with no previous fall offs available and no contraindications to DDAVP.

SUMMARY:
The Low Von Willebrand in Ireland Cohort (LoVIC) study focuses on the bleeding phenotype and biological mechanisms underlying low Von Willebrand Factor (VWF) levels.

DETAILED DESCRIPTION:
All patients with bleeding disorders in Ireland are registered on a national bleeding disorder database and attend the National Coagulation Centre in St. James's Hospital, Dublin, Ireland or the paediatric centre, Our Lady's Children's Hospital Crumlin for annual review. At review eligible patients will be invited to participate in the Low Von Willebrand in Ireland Cohort (LOVIC) study.

Following consent, an extensive bleeding assessment tool will be administered by a coagulation haematologist to all participants from which the International Society of Thrombosis and Haemostasis Bleeding Assessment Tool (ISTH BAT) and the Condensed Molecular and Clinical Markers for the Diagnosis and Management of Type 1 Von Willebrands Disease (MCMDM-1 VWD) scores can be derived. In addition, blood will be drawn for von Willebrand factor (VWF) measurements, VWF propeptide, platelet VWF. Citrated plasma and DNA will be stored for each patient. The relationship between laboratory parameters, (including von Willebrand factor, platelet VWF, FVIII and concomitant coagulation disorders) and the clinical phenotype in patients with low VWF will be studied. We will assess the effect of the laboratory parameters on the severity of bleeding tendency. In the future mutation analysis of the VWF gene will be performed in all participants in the LOVIC study.

Historical patient records and laboratory results will be reviewed and DDAVP (1-desamino-8-D-arginine vasopressin) fall off studies documented where available. If no previous DDAVP fall off study has been performed patients will be invited to attend.

ELIGIBILITY:
Inclusion Criteria:

* Two lowest VWF levels (VWF Antigen and/or VWF Ristocetin cofactor activity and/or VWF Collagen Binding) >30 IU/dL <50 IU/dL.

Exclusion Criteria:

* Pregnant patients
* Hospitalised patients/acutely unwell patients

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals (adults/children >3 years) with low Von Willebrand Factor (VWF) levels; defined as two lowest VWF levels (VWF Antigen and/or VWF Ristocetin cofactor activity and/or VWF Collagen Binding) >30 IU/dL <50 IU/dL.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-10; Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Number of Irish patients with Low Von Willebrand Factor with abnormal bleeding scores | at enrolment
  The ISTH-BAT and Condensed MCMDM-1 VWD score of all participants will be determined at enrollment using a physician directed questionnaire using only symptoms prior to their diagnosis with Low VWF. This will help elucidate the bleeding phenotype, if any, associated with Low VWF.

SECONDARY OUTCOMES:
The number of patients with Low VWF with abnormal plasma VWF clearance | 2 years
  For each individual enrolled the Von Willebrand factor propeptide (VWF:pp, U/dL), Von Willebrand factor antigen (VWF:Ag IU/dL) and Factor VIII:C (FVIII:C IU/dL) levels at enrolment will be determined. From this data the plasma VWF clearance will be ascertained using the plasma VWF:pp/VWF:Ag ratio. In addition, the FVIII:C/VWF:Ag ratio will be calculated to determine the contribution of altered VWF synthesis to Low VWF.
The rate of response to DDAVP in Irish patients with low Von Willebrand factor levels | 3 years
  For each individual with no contraindication a DDAVP trial will be performed with plasma VWF levels taken pre and at 1 and 4 hours post DDAVP. The rate of plasma VWF level fall off for each trial will be determined and the area under the curve (AUC) calculated. Complete response will be defined as a three fold increase from baseline.
The number of patients with Low VWF with reduced plasma VWF synthesis | 3 years
  For each individual enrolled the Von Willebrand factor antigen (VWF:Ag IU/dL) and Factor VIII:C (FVIII:C IU/dL) levels at enrolment will be determined. From this data the plasma FVIII:C/VWF:Ag ratio will be calculated to determine the contribution of altered VWF synthesis to Low VWF.

CONTACTS AND LOCATIONS:
Overall Officials: James S O'Donnell, MD,PhD, Principal Investigator — St. James's Hospital, Dublin Ireland
Locations (1):
- St. James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Doherty D, Michelle Lavin, Byrne M, Nolan M, O'Sullivan JM, Ryan K, O'Connell NM, Haberichter SL, Christopherson PA, Di Paola J, James PD, O'Donnell JS. Enhanced VWF clearance in low VWF pathogenesis: limitations of the VWFpp/VWF:Ag ratio and clinical significance. Blood Adv. 2023 Feb 14;7(3):302-308. doi: 10.1182/bloodadvances.2022007340. PMID 35523118
- [Derived] Aguila S, Lavin M, Dalton N, Patmore S, Chion A, Trahan GD, Jones KL, Keenan C, Brophy TM, O'Connell NM, Ryan K, Byrne M, Nolan M, Patel A, Preston RJS, James P, Di Paola J, O'Sullivan JM, O'Donnell JS. Increased galactose expression and enhanced clearance in patients with low von Willebrand factor. Blood. 2019 Apr 4;133(14):1585-1596. doi: 10.1182/blood-2018-09-874636. Epub 2019 Feb 15. PMID 30770394
- [Derived] Lavin M, Aguila S, Dalton N, Nolan M, Byrne M, Ryan K, White B, O'Connell NM, O'Sullivan JM, Di Paola J, James PD, O'Donnell JS. Significant gynecological bleeding in women with low von Willebrand factor levels. Blood Adv. 2018 Jul 24;2(14):1784-1791. doi: 10.1182/bloodadvances.2018017418. PMID 30042144
- [Derived] Lavin M, Aguila S, Schneppenheim S, Dalton N, Jones KL, O'Sullivan JM, O'Connell NM, Ryan K, White B, Byrne M, Rafferty M, Doyle MM, Nolan M, Preston RJS, Budde U, James P, Di Paola J, O'Donnell JS. Novel insights into the clinical phenotype and pathophysiology underlying low VWF levels. Blood. 2017 Nov 23;130(21):2344-2353. doi: 10.1182/blood-2017-05-786699. Epub 2017 Sep 15. PMID 28916584